CLINICAL TRIAL: NCT06595732
Title: Contin-RUN Study: Prevalence and Conservative Treatment of Urinary Incontinence in Female Runners
Brief Title: Contin-RUN Study: Urinary Incontinence in Female Runners
Acronym: Contin-RUN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Ana Paula Magalhães Resende, Clinical Professor Ana Paula M. Resende, PT, PhD, Principal Investigator, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 75069623.3.0000.5152
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; female runner; pelvic floor muscle training; Abdominal Hypopressive Technique
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1PFMT + Abd Group (Experimental): Participants in this group will perform pelvic floor muscle training in conjunction with abdominal muscle training. It is believed that abdominal contraction will lead to an increase in abdominal pressure, which will serve as additional load for pelvic floor muscle training.
  Interventions: Behavioral: Pelvic floor and abdominal training
- AHG Group (Experimental): Participants in this group will perform Hypopressive Abdominal Gymnastics exercises (Caufriez, 1997). It is believed that these exercises reduce the pressure on the pelvic floor muscles and help tone this musculature without causing harm.
  Interventions: Behavioral: Abdominal Hypopressive Technique Exercises
- PFMT Group (Active Comparator): Participants of PFMT group will perform specific exercises for the pelvic floor muscles, with maximum contraction and without involvement of other muscle groups. This arm is considered the control group because it is the treatment that has been proven to effectively treat urinary incontinence, as demonstrated in over 50 clinical trials.
  Interventions: Other: Pelvic floor muscle training

INTERVENTIONS:
Behavioral: Pelvic floor and abdominal training — Participants in this group will undergo 12 weeks of in-person training, with supervision by a specialist physical therapist, in groups of up to four women. The training will take place after an initial evaluation and will consist of 24 sessions, held twice a week. Exercises will target both the pelvic floor muscles and the abdominal muscles. The exercises will be divided into three phases, with progressively increasing difficulty each month. The progression will be achieved by increasing the load, the number of repetitions, and the complexity of the exercises.
  Arms: 1PFMT + Abd Group
Behavioral: Abdominal Hypopressive Technique Exercises — Participants in this group will perform Hypopressive Abdominal Gymnastics exercises as proposed by Marcel Caufriez (1997). The training will last 12 weeks and be conducted in person, with supervision by a specialist physical therapist, in groups of up to four women. The training will take place after an initial evaluation and will consist of 24 sessions, held twice a week. The exercises will be divided into three phases, with progressively increasing difficulty each month. Progression will be achieved by changing body positions, increasing the number of repetitions, and extending the duration of inspiratory apnea.
  Other Names: Hypopressive Exercises
  Arms: AHG Group
Other: Pelvic floor muscle training — Participants in this group will undergo 12 weeks of in-person training, supervised by a specialist physical therapist, in groups of up to four women. Specific exercises targeting the pelvic floor muscles will be performed, with voluntary and maximal contractions, without involving other muscle groups. The exercises will be divided into three phases, with progressively increasing difficulty each month. Progression will be achieved by increasing the load (transitioning from gravitational to antigravitational positions), increasing the number of repetitions, and combining sustained and rapid contractions to enhance the difficulty of execution.
  Arms: PFMT Group

SUMMARY:
This study comprises two phases, each with distinct objectives. The first phase aims to investigate the prevalence of urinary incontinence and other pelvic floor dysfunctions in Brazilian female runners through structured questionnaires. The second phase aims to evaluate and compare the effectiveness of three different exercise regimens for the treatment of urinary incontinence in female runners. The intervention groups include: a) pelvic floor muscle training combined with abdominal training, b) hypopressive abdominal exercises, and c) pelvic floor muscle training alone. The primary outcome measure is the severity of urinary incontinence, which will be assessed using the adapted 1-hour pad test and a 3-day bladder diary. Secondary outcomes include symptoms of pelvic floor dysfunction and pelvic floor muscle function. The intervention will last for 12 weeks, after which participants will be reassessed to determine which training regimen is most effective in treating urinary incontinence in female runners.

DETAILED DESCRIPTION:
This study has two stages with distinct objectives. The first stage aims to investigate the prevalence of urinary incontinence and other pelvic floor dysfunctions in Brazilian female runners. To achieve this goal, a survey will be conducted using a questionnaire, which will include questions about demographic data, general gynecological and obstetric health (menopause, pregnancies, deliveries), training specifics (weekly volume, time spent running, practice of other exercises, how the training is conducted), and questions related to pelvic floor dysfunctions (urinary incontinence, fecal incontinence, sexual dysfunctions, and symptoms of genital prolapse). For this study, it is estimated that at least 400 female runners will respond to the questionnaire.

The second stage aims to compare three types of exercise programs for the treatment of urinary incontinence in runners: (1) pelvic floor muscle training combined with abdominal training; (2) hypopressive abdominal gymnastics; or (3) pelvic floor muscle training. The primary outcome of interest is the severity of urinary loss, assessed by a 1-hour adapted pad test and a 3-day voiding diary. Secondary outcomes will include symptoms related to urinary incontinence and other dysfunctions. For this purpose, the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) and Pelvic Floor Distress Inventory (PFDI-20) will be used. Lastly, pelvic floor muscle function will be assessed through vaginal palpation, quantified using the Oxford scale, and through vaginal manometry. After agreeing to participate and signing the informed consent form, the women will be evaluated and then randomized into one of the three previously described groups. The exercises will be performed over a 12-week period. The women will then be re-evaluated. A sample size calculation was performed, and 58 participants will be required in each group to verify the superiority of one type of exercise over the others.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been running for at least six months
* Run at least 15 kilometers per week,
* Have no injuries that have prevented them from running for more than three weeks in the past six months
* Experience involuntary urinary leakage during running
* The women must have a pelvic floor muscle strength of ≥ 2 on the modified Oxford scale

Exclusion Criteria:

* Having a diagnosed neuromuscular disease that affects bladder function
* Having undergone previous pelvic or perineal surgeries for the correction of pelvic floor dysfunctions
* Having previously received physical therapy for the treatment of pelvic floor dysfunctions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals assigned female at birth, who have a vagina, who are runners, and who experience urinary leakage during running.
Enrollment: 174 (Estimated)
Dates: Start 2023-08-03 (Actual); Primary Completion 2025-06-17 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
Amount of urinary leakage during running | From enrollment to the end of the treatment at 12 weeks
  The severity of urinary incontinence is the primary outcome of interest. The amount of urinary leakage will be assessed using a modified 1-hour pad test.
  The pad test will be performed on a treadmill. The participant will drink 500 ml of water in 15 minutes, wait another 15 minutes in rest, place a pre-weighed pad in her underwear, and then run continuously for 40 minutes on the treadmill at a comfortable speed of her choice. After the running period, the pad will be removed and weighed to determine the amount of urinary leakage in grams.

SECONDARY OUTCOMES:
Frequency of urinary leakage | From enrollment to the end of the treatment at 12 weeks
  The frequency of urinary leakage will be evaluated through a bladder diary. The bladder diary will be completed over three days, during which the participant will record daytime urinary frequency, nighttime urinary frequency, the number of urinary leakage episodes, and the number of pad changes (if that's the case). The information will be logged for three consecutive days, and the participant will be required to run on at least two of those days.
Other pelvic floor dysfunction symptoms | From enrollment to the end of the treatment at 12 weeks
  In order to achieve this outcome, The Pelvic Floor Distress Inventory (PFDI-20) will be used. This is a self-administered quality of life questionnaire containing 20 questions that assess whether the individual has specific symptoms related to the bowel, bladder, or pelvis. If they do, they must rate how bothersome these symptoms are. Scores range from 0 to 100, the higher the score, the greater the discomfort in woman's life.
Pelvic floor muscle strength | From enrollment to the end of the treatment at 12 weeks
  Pelvic floor muscle strength will be assessed through vaginal palpation. Palpation will be performed to measure the strength of the pelvic floor muscles using the modified 0-5 Oxford scale.
Pelvic floor manometry | From enrollment to the end of the treatment at 12 weeks
  The vaginal squeeze pressure of the pelvic floor muscles will be assessed through manometry. The Peritron manometer will be used to measure peak pressure and the average pressure exerted by the contraction of the pelvic floor muscles.
Impact of urinary incontinence in the quality of life | From enrollment to the end of the treatment at 12 weeks
  The impact of urinary incontinence on quality of life will be the secondary outcome of interest. To assess this impact, the authors are going to use the International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF). It is a self-administered tool consisting of four questions that evaluate the frequency, severity, and impact of urinary incontinence, in addition to a set of eight self-diagnosis items related to the causes or situations of urinary incontinence experienced by women. The overall score is obtained by summing the scores from questions 3, 4, and 5, and the higher the value, the worse the quality of life and the more the symptom affects the individual's life.

CONTACTS AND LOCATIONS:
Locations (1):
- Benjamin Constant St, 1286, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
After data collection, the research team will meet to decide whether to share individual evaluation data, while ensuring that participants are not identified for ethical reasons. Spreadsheets containing data on outcomes for each individual, as well as other information such as age, body mass index, menopause status, etc., may be shared to facilitate the development of systematic reviews and meta-analyses on the topic. This would benefit the entire scientific and academic community, and ultimately the general population, as understanding the best treatment evidence helps individuals receive more targeted and effective treatment.